CLINICAL TRIAL: NCT03105843
Title: Sensory-Mechanical Responses to Eucapneic Voluntary Hyperventilation and Mannitol in Individuals With Cough Variant Asthma and Chronic Cough
Brief Title: Sensory-Mechanical Responses to Eucapneic Voluntary Hyperventilation and Mannitol
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Diane Lougheed (Other)
Responsible Party: Sponsor-Investigator, Dr. Diane Lougheed, Professor of Medicine, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-17
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Asthma; Cough; Cough Variant Asthma
Keywords: Asthma; Cough; Eucapneic Voluntary Hyperventilation; Hypertonic Saline
MeSH Terms: conditions — Asthma; Cough; Cough-Variant Asthma | interventions — Methacholine Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cough Variant Asthma (Experimental): Individuals diagnosed with Cough variant asthma
  Interventions: Drug: Methacholine (MCh) Challenge Testing; Diagnostic Test: Eucapneic Voluntary Hyperventilation (EVH); Drug: Mannitol Inhalation Kit
- Methacholine-induced cough (Experimental): Individuals with chronic cough and negative methacholine challenge
  Interventions: Drug: Methacholine (MCh) Challenge Testing; Diagnostic Test: Eucapneic Voluntary Hyperventilation (EVH); Drug: Mannitol Inhalation Kit
- Control (Experimental): Individuals with no history of asthma or chronic cough
  Interventions: Drug: Methacholine (MCh) Challenge Testing; Diagnostic Test: Eucapneic Voluntary Hyperventilation (EVH); Drug: Mannitol Inhalation Kit

INTERVENTIONS:
Drug: Methacholine (MCh) Challenge Testing — Visit 1: Informed consent, Baseline screening and pulmonary function tests and Low-dose methacholine challenge testing using partial and full flow-volume loops.
  Other Names: MCh[inhalation of sequential doubling doses of MCh(0.0625-16 mg/mL)]; Provocholine
Diagnostic Test: Eucapneic Voluntary Hyperventilation (EVH) — Visit 2 or 3: Will be conducted in random order and subjects will perform one of the two challenge tests at either visit.
Drug: Mannitol Inhalation Kit — Visit 2 or 3: Will be conducted in random order and subjects will perform one of the two challenge tests at either visit.
  Other Names: Mannitol Challenge Test

SUMMARY:
The objectives of this study are to determine the sensory-mechanical responses to Eucapneic Voluntary Hyperventilation (EVH) and Mannitol in individuals with cough variant asthma (CVA) and methacholine-induced cough with normal airway sensitivity (COUGH) and compare these responses to a control group of healthy individuals without asthma or chronic cough.

We hypothesize:

1. EVH and Mannitol cause dyspnea, cough, small airway obstruction with resultant dynamic hyperinflation, gas trapping and autoPEEP in individuals with CVA and COUGH, but not healthy controls.
2. The sensory-mechanical responses to both hyperosmolar challenges (EVH and Mannitol) are comparable within groups (CVA, COUGH and healthy controls).

DETAILED DESCRIPTION:
Asthma is a chronic respiratory condition characterized by eosinophilic airway inflammation. Individuals with classic asthma experience paroxysmal symptoms including cough, wheeze, shortness of breath and chest tightness. Cough variant asthma (CVA) is asthma in which chronic cough (cough lasting eight weeks or more) is the sole or predominant symptom of asthma. The pathophysiologic mechanisms which differentiate asthma, CVA, and eosinophilic bronchitis without asthma are not fully understood. We have recently identified individuals with chronic cough who cough during methacholine but have normal airway sensitivity (ie. do not have asthma or CVA) (COUGH) and may or may not have eosinophilic bronchitis. The purpose of this research is to further explore the pathophysiologic basis for cough in these conditions using two 'indirect' inhalation challenge tests: eucapneic voluntary hyperventilation (EVH) and Mannitol), which induce osmotic and/or temperature changes in airway. Specifically, this study will collect preliminary data on the sensory-mechanical responses of individuals with CVA, COUGH and healthy controls to EVH and Mannitol Challenges.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65 years of age with CVA and individuals with methacholine-induced cough but normal airway sensitivity. The following definitions will be used:

  1. CVA: chronic cough (≥8 weeks) is the sole or predominant symptom and positive methacholine challenge (PC20 ≤ 16 mg/mL) and history of cough responding to specific asthma treatment (such as inhaled steroid or 1 week trial of bronchodilator);
  2. Methacholine-induced cough but normal airway sensitivity: chronic cough (≥8 weeks) is the sole or predominant symptom and negative methacholine challenges (PC20 > 16 mg/mL).
* Individuals aged 18-65 years of age with no history of asthma or chronic cough.

Exclusion Criteria:

* an exacerbation necessitating a change in medication, emergency department visit or hospitalizations within the previous 4 weeks
* inability to perform acceptable spirometry
* medical contraindications to methacholine challenge testing
* smoking history in excess of 10 pack years Note: Previous treatment with inhaled or systemic corticosteroids is not an exclusion criterion; medication use will be recorded and examined in the analysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mid expiratory flows | Time frame of the methacholine challenge varies between individuals. At provocative dose/ventilation causing a 20% decline in FEV1 (PD20 and PC20 respectively). On average, these occur about 15-25 minutes into the challenge test
  The bronchodilating effect of a DI will be examined using responses to the challenge testing (Visit 2/3) in these subgroups by comparing the mid-expiratory flow difference between the partial (PEF) and full maximal flow-volume (MEF) loops at 40% above Residual Volume (RV) from the forced vital capacity (FVC) (PEF40 and MEF40 respectively) at provocative dose of 4.5% saline causing a 20% decline in FEV1 (PD20 (HS)) and provocative minute ventilation causing a 20% decline in FEV1 (PC20 (EVH)) with that recorded at baseline.

SECONDARY OUTCOMES:
Respiratory System Reactance (X5) | After dose administration; will occur 2-5 minutes after dose
  Single IOS will measure peripheral airway function using respiratory system reactance (X5) and peripheral resistance (R5-R20) and central resistance (R20) will be used as an index of airway narrowing.
Peripheral Resistance (R5-R20) | After dose administration; will occur 2-5 minutes after dose
  Single IOS will measure peripheral airway function using respiratory system reactance (X5) and peripheral resistance (R5-R20) and central resistance (R20) will be used as an index of airway narrowing.
Central Airway Resistance | After dose administration; will occur 2-5 minutes after dose
  Single IOS will measure peripheral airway function using respiratory system reactance (X5) and peripheral resistance (R5-R20) and central resistance (R20) will be used as an index of airway narrowing.
Forced Vital Capacity (FVC) | After dose administration; will occur 2-5 minutes after dose
  As an index of airway closure.
FEV1/FVC | After dose administration; will occur 2-5 minutes after dose
  As an index of airway obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: M. Diane Lougheed, MD, MSc, Principal Investigator — Department of Medicine, Queen's University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No